CLINICAL TRIAL: NCT06759662
Title: Association of Neutrophil- Lymphocyte Count Ratio and Microbial Infection in Hospitalized Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Hamed Abdelwahed Mohamed, residant doctor at Assiut university hospital, Assiut University
Other Study IDs: N-L count ratio microbial inf
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Microbial Infection
Keywords: neutrophil- lymphocyte count ratio

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- microbial infections cases: All cases diagnosed with microbial infections at Assiut university hospitals

SUMMARY:
Microbial infection is one of leading cause of morbidity and mortality in the world. Bacteremia that result from microbial infection has mortality rate as high as 30% . Systemic infections that result from microbial infection is a generalized disease that progresses rapidly and can lead to high mortality. This infection sets in from a progression of various pathogenic microorganisms that enter the bloodstream, reproduce and then release toxins and metabolites . Early diagnosis of microbial infection is essential for treatment. Culturing microorganisms is the most definitive way to confirm bacterial infections. Unfortunately, this gold standard is time consuming and may take from 24 to 48 hours and sometimes up to a week. A number of rapid initial indicators of microbial infection have been proposed, including C-reactive protein, neutrophil count, and white blood cell count. However, these criteria do not always reliably distinguish between severe bacterial, fungal, and viral infections . Therefore, the neutrophil-to-lymphocyte ratio (NLCR), a simple ratio between the number of neutrophils and lymphocytes measured in peripheral blood, has been proposed as a biomarker that combines two aspects of the immune system: the innate immune response, which is mainly driven by neutrophils, and adaptive immunity, supported by lymphocytes . This study aims to determine the diagnostic value of the neutrophil-to-lymphocyte ratio (NLCR) as an indicator of microbial infection, using complete blood count to determine the ratio in addition to culture and sensitivity according to the site of infection.

the aim of this study is to Investigating the association between neutrophil-lymphocyte count and the presence of microbial infection in the hospitalized patients.

DETAILED DESCRIPTION:
Microbial infection is one of leading cause of morbidity and mortality in the world. Bacteremia that result from microbial infection has mortality rate as high as 30% . Systemic infections that result from microbial infection is a generalized disease that progresses rapidly and can lead to high mortality. This infection sets in from a progression of various pathogenic microorganisms that enter the bloodstream, reproduce and then release toxins and metabolites . Early diagnosis of microbial infection is essential for treatment. Culturing microorganisms is the most definitive way to confirm bacterial infections. Unfortunately, this gold standard is time consuming and may take from 24 to 48 hours and sometimes up to a week. A number of rapid initial indicators of microbial infection have been proposed, including C-reactive protein, neutrophil count, and white blood cell count. However, these criteria do not always reliably distinguish between severe bacterial, fungal, and viral infections . Therefore, the neutrophil-to-lymphocyte ratio (NLCR), a simple ratio between the number of neutrophils and lymphocytes measured in peripheral blood, has been proposed as a biomarker that combines two aspects of the immune system: the innate immune response, which is mainly driven by neutrophils, and adaptive immunity, supported by lymphocytes . This study aims to determine the diagnostic value of the neutrophil-to-lymphocyte ratio (NLCR) as an indicator of microbial infection, using complete blood count to determine the ratio in addition to culture and sensitivity according to the site of infection.

ELIGIBILITY:
Inclusion Criteria:

* age more than 18 years old
* both sex
* conformed diagnosis with micorbial infection

Exclusion Criteria:

* Immunodeficiency patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All cases diagnosed with microbial infections at Assiut university hospitals.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
neutrophil-lymphocyte count ratio | baseline
  neutrophil-lymphocyte count ratio in the hospitalized patients with microbial infection

IPD SHARING:
Plan to Share IPD: Undecided